CLINICAL TRIAL: NCT05116111
Title: A Randomized, Multi-center, Double-blind, Parallel-group, Placebo-controlled Phase II Study To Evaluate the Safety, Tolerance, Pharmacokinetics/Pharmacodynamics and Efficacy of SYHA1402 Tablets For the Treatment of Patients With Diabetic Peripheral Neuropathy in China
Brief Title: A Study To Evaluate the Safety, Tolerance, Pharmacokinetics/Pharmacodynamics and Efficacy of SYHA1402 Tablets For the Treatment of Patients With Diabetic Peripheral Neuropathy in China
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HA1403-CSP-004
Record Dates: First submitted 2021-09-03; First posted 2021-11-10 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Distal Symmetric Polyneuropathy (DSPN)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SYHA1402 1000 mg plus placebo 500 mg (Experimental): Eligible patients will be randomly assigned to receive SYHA1402 1000 mg and placebo 500 mg twice daily for 16 weeks of treatment after a placebo introduction period.
  Interventions: Drug: SYHA1402 tablets; Drug: Placebo
- SYHA1402 1500 mg (Experimental): Eligible patients will be randomly assigned to receive SYHA1402 1500 mg twice daily for 16 weeks of treatment after a placebo introduction period.
  Interventions: Drug: SYHA1402 tablets
- Placebo 1500 mg (Placebo Comparator): Eligible patients will be randomly assigned to receive placebo 1500 mg twice daily for 16 weeks of treatment after a placebo introduction period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SYHA1402 tablets — SYHA1402 tablets, oral, twice daily
  Arms: SYHA1402 1000 mg plus placebo 500 mg; SYHA1402 1500 mg
Drug: Placebo — Placebo, oral, twice daily
  Arms: Placebo 1500 mg; SYHA1402 1000 mg plus placebo 500 mg

SUMMARY:
This study aims to evaluate the safety, tolerance, pharmacokinetics/pharmacodynamics and efficacy of SYHA1402 tablets for the treatment of patients with diabetic peripheral neuropathy (DPN) in China.

DETAILED DESCRIPTION:
This is a randomized, multi-center, double-blind, parallel-group, placebo-controlled, phase II clinical trial to evaluate safety, tolerance, pharmacokinetics/pharmacodynamics and efficacy of SYHA1402 tablets in DPN patients. A total number of 135 patients will be randomized (2:2:1) into three groups. Patients between 18 and 75 years old and diagnosed with a Distal Symmetric Polyneuropathy (DSPN) prior to study enrolment will be enrolled. The study consists of 4 stages: a 2-week screening period, a 1-week placebo introduction period, a 16-week randomized double-blind treatment period, and a 2-week post-study follow-up period. The overall planned duration of this study is approximately 21 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained before any trial-related activities voluntarily, understanding the procedures and methods of this study, and be willing to strictly follow the trial protocol;
2. Males or females, aged 18-75 years (both inclusive);
3. Diagnosed with type 1 or type 2 diabetes for more than 6 months, hemoglobin Alc (HbA1c) between 7% and 10% at screening, fasting plasma glucose (FPG) <11.1 mmol/L, and the glucose-lowering treatment has been stable for at least 30 days and is expected to remain unchanged throughout the study;
4. According to the 《China Type 2 Diabetes Prevention and Cure Guidelines (2020 edition)》, those diagnosed with diabetic peripheral neuropathy are classified as distal symmetric polyneuropathy (DSPN), the diagnostic criteria consists of:(1) A clear history of diabetes; (2) Neuropathy appeared during or after diagnosis of diabetes; (3) Symptoms and signs are consistent with the performance of DPN; (4) Patients with clinical symptoms (pain, numbness, abnormal sensation, etc.), with abnormality in any 1 of 5 examinations (ankle reflexes, needle pain, vibration, pressure, temperature); Patients without symptoms, with abnormalities in any 2 of 5 examinations and a clinical diagnosis of DPN; (5) Excluding patients with neuropathy caused by other causes;
5. Toronto Clinical Neuropathy Score (TCNS) ≥ 6 points, with sensory test score ≥ 2 points at screening and baseline.

Exclusion Criteria:

Those who meet any of the exclusion criteria will not be enrolled:

1. Patients with peripheral neuropathy caused by other diseases: such as cervical and lumbar vertebral disease, cerebrovascular disease, intracranial tumor or trauma, toxic peripheral neuropathy (e.g. chemotherapy, alcohol), Guillain-Barr é syndrome, multiple sclerosis, bone joints or tendon lesions, severe arteriovenous and vascular lesions, severe liver and kidney insufficiency, hyperthyroidism or degeneration, subclinical thyroid dysfunction, vitamin B12 deficiency, infection (e.g. human immunodeficiency virus), etc;
2. Patients with previous peripheral arterial disease, and significant intermittent claudication symptoms or previous lower extremity vascular bypass or angioplasty at screening;
3. History of malignant neoplasms (except cured basal cell skin cancer, in-situ carcinomas and papillary thyroid cancer) or history of antineoplastic therapy within 5 years prior to screening;
4. Patients with a change of more than 2 points in the same item of the mTCNS at screening and baseline;
5. Visual Analogue Scale (VAS) > 8 points at screening;
6. Diabetic foot, diabetic peripheral vascular lesions, lower limb amputation, diabetic muscular atrophy, Charcot joint disease within 3 months prior to screening;
7. Acute complications such as severe hypoglycemia with loss of consciousness, diabetic ketoacidosis, diabetic hyperosmolar hyperglycemia syndrome, lactic acidosis, etc. within 3 months prior to screening;
8. Those who have used a prohibited combination drug within 3 months before screening must discontinue the drug for at least 1 month or 5 half-lives (whichever is longer) prior to screening visit, and the drug must be discontinued throughout the study period;
9. Any of the following cardiovascular events within 6 months prior to screening: unstable angina requiring hospitalization, myocardial infarction, coronary artery bypass transplantation, transdermal coronary intervention (diagnostic angiography is permitted), moderate to severe congestive heart failure (NYHA III or IV), atrial or ventricular arrhythmia (e.g. atrial fibrillation, ventricular tachycardia, etc.) requiring hospitalization, pacemaker or defibrillator implantation, temporary cerebral ischemic attacks or cerebrovascular accidents (e.g. strokes); Or coronary artery bypass grafting or revascularization is planned during the study;
10. Uncontrolled severe hypertension (untreated or post-treated) at screening, defined as systolic blood pressure ≥160 mm Hg or diastolic blood pressure ≥100 mm Hg;
11. Those who with awake pulse < 60 BPM or > 100 BPM at screening；
12. The Body Mass Index (BMI) < 18.5 kg/m^2 or > 35 kg/m^2 at screening, calculated by BMI = body weight (kg)/height^2(m^2);
13. Grade II or III atrioventricular block occurred in 12-lead ECG (in the absence of a pacemaker) at screening, long QT syndrome or QTc > 450 ms (male) / 470 ms (female);
14. Any active infections at screening, including but not limited to urinary tract infections, upper respiratory tract infections, diabetic foot infections, etc., and who needs further treatment;
15. Severe hematologic, hepatic, or renal abnormalities at screening with any laboratory assessments meeting the following criteria: 1)Platelet count < 100 × 10^9/L; 2) Aspartate Aminotransferase (AST) or alanine aminotransferase (ALT) ≥ 2.5 × upper limit of normal (ULN) of the reference range, or total bilirubin ≥ 1.5 × ULN of the reference range; 3) Creatine kinase > 2.0 × ULN; 4) Estimated renal glomerular Filtration Rate (eGFR) < 60 mL/(min*1.73m^2) (calculated using the CKD-EPI formula); 5) Triglycerides (TG) > 5.6 mmol/L;
16. HBsAg-positive with HBV DNA copy number above the lower limit of the HBV DNA test, or HCV antibodies (HCV Ab)-positive with HCV RNA copy number above the lower limit of the HCV RNA test, human immunodeficiency virus antibody (HIV Ab) positive, serum syphilis helix antibody (TP Ab) positive with syphilis helix titrating positive at screening;
17. Thyroid dysfunction (FT3, FT4, TSH examination with clinically significant abnormalities) at screening, including undergoing treatment;
18. Cannot swallow oral drugs, or suffer from diseases that affect oral drug absorption, distribution, metabolism, excretion, as well as diseases that affect the evaluation of the efficacy and safety of experimental drugs, such as active bowel disease, partial or complete intestinal obstruction, chronic diarrhea, etc;
19. Patients who are allergic to any ingredient in the test drug;
20. Patients with severe bleeding disorders;
21. Conditions that may affect the evaluation of efficacy, such as skin diseases in the affected skin area that may affect the evaluation of nerve conduction function;
22. Pregnancy, breast-feeding, the intention of becoming pregnant during the trial; or women of childbearing potential (WOCBP) or male patient do not wish to use adequate contraceptive measures from the time signing the informed consent form until 3 months after the last dose of the study drug;
23. Patients who have a history of alcohol addiction or substance abuse prior to screening (alcohol addiction is defined as regular daily alcohol consumption in excess of the following standard amounts: 720 mL of beer, 300 mL of red wine or 90 mL of liquor, approximately 20 g of alcohol) or an inability to limit alcohol consumption to this standard throughout the study period;
24. Patients who have smoked more than 10 cigarettes (including 10 cigarettes) per day in the three months before screening or who could not control less than 10 cigarettes per day during the whole study period;
25. Participation in other trials within 3 months prior to screening;
26. Risk of incompliance and/or inability to complete the trial, as judged by the investigator, including but not limited to: psychiatric disorder (such as eating disorder), mental incapacity, unwillingness or evidence of uncooperative attitude, language barriers precluding adequate understanding of the trial (including inability to read or write);
27. Patient compliance < 80% or > 120% during the introductory period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2021-12-31 (Estimated); Primary Completion 2023-05-15 (Estimated); Study Completion 2023-06-15 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in modified Toronto Clinical Neuropathy Score (mTCNS)- Sensory Test Score at week 16 | From baseline to week 16 post-dose
  To Compare SYHA1402 with placebo, the overall score and symptom score of mTCNS changes from baseline at week 16. The mTCNS examines signs and symptoms of polyneuropathy. It consists of a questionnaire which explores the presence of foot pain, numbness, tingling, weakness, and loss of sensation leading to ataxia. Secondly, sensory tests will be performed including sensation for pinprick, light touch, temperature, vibration and position sense. The minimum value is 0 meaning the patient does not show any signs or symptoms of polyneuropathy and the maximum value is 33 meaning the patient presents with severe signs and symptoms of polyneuropathy.

SECONDARY OUTCOMES:
Change from baseline in overall score and symptom score of mTCNS at week 16 | From baseline to week 16 post-dose
  To Compare SYHA1402 with placebo, the overall score and symptom score of mTCNS changes from baseline at week 16. The mTCNS examines signs and symptoms of polyneuropathy. It consists of a questionnaire which explores the presence of foot pain, numbness, tingling, weakness, and loss of sensation leading to ataxia. Secondly, sensory tests will be performed including sensation for pinprick, light touch, temperature, vibration and position sense. The minimum value is 0 meaning the patient does not show any signs or symptoms of polyneuropathy and the maximum value is 33 meaning the patient presents with severe signs and symptoms of polyneuropathy.
Change from baseline in Toronto Clinical Neuropathy Score (TCNS) at week 16 | From baseline to week 16 post-dose
  To Compare SYHA1402 with placebo, the Toronto Clinical Neuropathy Score (TCNS) changes from baseline at week 16. Scales are defined as follows: 0-5 = no neuropathy; 6-8 = mild neuropathy; 9-11 = moderate neuropathy; ≥ 12 = severe neuropathy.
Change from baseline in Nerve Conduction Velocities (NCVs) and Amplitude at week 16 | From baseline to week 16 post-dose
  To Compare SYHA1402 with placebo, the Nerve Conduction Velocities (NCVs) and Amplitude changes from baseline at week 16.
Change from baseline in Visual Analogue Scale (VAS) at week 16 | From baseline to week 16 post-dose
  To Compare SYHA1402 with placebo, the Visual Analogue Scale (VAS) changes from baseline at week 16. Including local pain, limb numbness, paresthesia (e.g. burning sensation, formication, electrical sensation). Participants rated their pain on a 100 millimeter (mm) Visual Analog Scale (VAS) ranging from 0 mm = no pain to 100 mm = worst possible pain.
Change from baseline in the 36-Item Shot-Form Health Survey (SF-36) score at week 16 | From baseline to week 16 post-dose
  To Compare SYHA1402 with placebo, the 36-Item Shot-Form Health Survey (SF-36) score changes from baseline at week 16. The SF-36 quality of life scale is used to monitor change in subject reported functionality, well-being, and overall health status. The score of each part ranges from 0 (worst score) to 100 (best score).
Clearance (CL) | Pre-dose and multiple timepoints up to 16 weeks
  Rate and Extent of Absorption SYHA1402 by Assessment of the Apparent Clearance
Volume of Distribution (V) | Pre-dose and multiple timepoints up to 16 weeks
  Rate and Extent of Absorption SYHA1402 by Assessment of the Apparent Volume of Distribution
Pharmacodynamics (PD) indicator | Pre-dose and multiple timepoints up to 16 weeks
  Proportional change from baseline in whole blood/red blood cell sorbitol concentration (%)
Incidence of adverse events (AEs) | Throughout the study period, an average of 21 weeks
  Incidence of adverse events (AEs)

IPD SHARING:
Plan to Share IPD: Undecided